CLINICAL TRIAL: NCT00556244
Title: Pars Plana Vitrectomy for Diabetic Fibrovascular Proliferation With and Without Internal Limiting Membrane Peeling
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 200704053M
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-04

CONDITIONS: Patients With Proliferative Diabetic Retinopathy Who Have Active Fibrovascular Proliferation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Active Comparator)
  Interventions: Procedure: ILM peeling

INTERVENTIONS:
Procedure: ILM peeling — ILM maculorhexis is initiated using scraper and completed using a 25-gauge Synergetics (St. Louis, MO) forceps.

SUMMARY:
Internal limiting membrane peeling in diabetic vitrectomy will help prevent postoperative epiretinal membrane formation

DETAILED DESCRIPTION:
Progressive fibrovascular proliferation may occur despite appropriate panretinal photocoagulation in diabetic patients. Fibrovascular proliferation may lead to persistent or recurrent vitreous hemorrhage, macular traction, or traction macular detachment, and becomes a major indication for vitrectomy.1 During the past 25 years, anatomical and visual results of vitrectomy for severe proliferative diabetic retinopathy have improved as a result of improved understanding of the pathoanatomy and improvements in surgical instrumentation.2-5 Although anatomical success is high after complete vitrectomy, recurrent epiretinal membrane may cause macular thickening, cysts formation, preventing good functional outcome.6 An epiretinal membrane (ERM) is a non-vascular cellular membrane that may cause symptomatic visual disturbances due to retinal wrinkling and distortion.7 These epiretinal membranes have been found to be composed of fibroblasts, glial cells, macrophages, myofiboblasts, nad retinal pigment epithelial cells.8-9 Studies have suggested removal of internal limiting membrane (ILM) may decrease the likelihood of post-operative ERM formation in cases of diabetic macular edema and idiopathic ERM. It is postulated that removal of the ILM removes the scaffold upon which myofibroblasts would proliferate.10 Efficacy of vitrectomy including removal of ILM was mostly described as facilitating resolution of diffuse diabetic macular edema11 and improvement of visual acuity or in macular hole surgery in diabetic patients.12However, it is unknown if removal of ILM during vitreoretinal surgery in diabetic patients with active fibrovascular proliferation is useful in preventing postoperative ERM formation. The purpose of this study is to compare the postoperative epiretinal membrane (ERM) formation and visual outcome in diabetic patients with active fibrovascular proliferation who underwent vitrectomy with or without ILM peeling.

ELIGIBILITY:
Inclusion Criteria:

* active fibrovascular proliferation with or without tractional detachment
* previous pan-retinal photocoagulation at least 3 months before

Exclusion Criteria:

* biomicroscopic evidence of macular hole
* combination of tractional and rhegmatogenous retinal detachment
* location of fibrovascular proliferation anterior to the equator
* major ocular surgery history(including, scleral buckle, glaucoma filter, cornea transplant, vitreoretinal surgery etc
* the presence of other ocular conditions such as glaucoma, uveitis, or other ocular inflammatory diseases.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Study Completion 2007-11 (Estimated)

PRIMARY OUTCOMES:
Snellen BCVA and epiretinal membrane formation measured with OCT | within 6 months after the surgery

SECONDARY OUTCOMES:
central macular thickness measured bt OCT | within 6 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chung-may Yang, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan